CLINICAL TRIAL: NCT01825291
Title: Sleep-disordered Breathing in Postmenopausal Women and CPAP Treatment
Brief Title: Sleep-disordered Breathing in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1/2000
Record Dates: First submitted 2013-02-22; First posted 2013-04-05 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; co-morbidities of sleep apnea; CPAP treatment
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- sleep apnea
  Interventions: Procedure: CPAP treatment

INTERVENTIONS:
Procedure: CPAP treatment

SUMMARY:
The purpose of this study is to investigate the effectiveness of CPAP treatment to co-morbidities of sleep apnea by looking the change of the consumption of medication of the co-morbidities before and after starting the CPAP treatment.

DETAILED DESCRIPTION:
Sleep-disordered breathing (SDB) is frequently linked with cardiovascular diseases including stroke and type 2 diabetes, which increase the indirect costs of sleep apnea. Also non-cardiovascular co-morbidities are possible but seldom studied. CPAP treatment reverses the increased healthcare utilization seen before the sleep apnea diagnosis.

Previous studies addressing the cardiovascular co-morbidities in SDB have focused on obstructive sleep apnea and in male populations, but not on partial upper airway obstruction. Partial upper airway obstruction is common in both genders but especially in women. According to investigators' clinical experience, women with partial upper airway obstruction are especially likely to have severe symptoms from their SDB. There are scarce data on cardiovascular co-morbidities associated with partial upper airway obstruction and the female gender.

To study the prevalence of co-morbidities adding to the burden of SDB (periodic obstructive breathing and partial upper airway obstruction), investigators applied a conservative but robust strategy using the governmental database of medication reimbursed by the public health insurance system. Investigators analyzed both the cardiovascular and non-cardiovascular co-morbidities in our clinical population of SDB, separately in patients with periodic obstructive breathing or with partial upper airway obstruction during sleep.Investigators found that concomitant diseases ware common in SDB. Asthma and/or COPD were surprisingly frequent, and also chronic hypertension had an increased prevalence. In addition, males had diabetes mellitus and females hypothyroidism more than general population. The results emphasize the importance of diagnosis and treatment of the co-morbidities such as asthma, COPD, hypertension, diabetes and thyroid insufficiency regardless if the patient has partial upper airway obstruction or obstructive sleep apnea.

Now, investigators hypothesize that CPAP treatment reduces the consumption of medication of the co-morbidities of sleep apnea. Therefore, a retrospective analyze of 5 year before and 5 year after starting the CPAP treatment the medication consumption of the same population previously used will be conducted. To do this, the governmental database of medication reimbursed by the public health insurance system will be used.

ELIGIBILITY:
Inclusion Criteria:

* patient with sleep apnea
* CPAP treatment started and continued

Exclusion Criteria:

* no CPAP treatment started

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical sample of patients with sleep apnea
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1999-01; Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the consumption of medication of co-morbidities of sleep apnea | 5 year before CPAP treatment and 5 year after CPAP treatment
  The amount of medication used gathered from the National Agency for Medicines and Social Insurance Institution database.